CLINICAL TRIAL: NCT06371716
Title: Application of a New System of Ultrasound (US) Guided - Radiofrequency Ablation (RFA) on Explanted Pancreas From Patients With Solid Pancreatic Masses: Study of Efficacy
Brief Title: Ex-vivo Ultrasound Guided Radiofrequency Ablation on Pancreatic Solid Lesions
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: resectable pancreatic adenocarcinoma and neuroendocrine pancreatic neoplasms are difficult to be enrolled. Pancreatic resectable cancers are treated nowadays with chemotherapy and big neuroedocrine pancreatic lesions rare
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Paolo Giorgio Arcidiacono, MD, Professor, IRCCS San Raffaele
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EUS-RFA ex-vivo 2016
Record Dates: First submitted 2024-03-25; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Pancreatic Cancer; Endoscopic Ultrasound; Radiofrequency Ablation
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: 15 resected PDAC without neoadjuvant treatment 15 resected PDAC with neoadjuvant treatment 15 resected neuroendocrine tumors
  Each group (15 patients each) Subgroup A: 10 W (5 patients) Subgroup B: 30 W (5 patients) Subgroup C: 50 W (5 patients)
Who Masked: Participant, Outcomes Assessor
Masking Description: pathologists (two different pathologist blinded about the power of RFA applied and respect to the other pathologist) will evaluate the effect of ablation (coagulative necrosis at microscopic evaluation)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- resected PDAC without neoadjuvant chemotherapy treatment (Experimental): Subgroup A: 10 W (5 patients) Subgroup B: 30 W (5 patients) Subgroup C: 50 W (5 patients)
  Interventions: Procedure: ex-vivo RFA under US control at 10 Watts (W) of power in 3 differents arms of lesions; Procedure: ex-vivo RFA under US control at 30 Watts (W) of power in 3 differents arms of lesions; Procedure: ex-vivo RFA under US control at 50 Watts (W) of power in 3 differents arms of lesions
- resected PDAC with neoadjuvant chemotherapy treatment (Experimental): Subgroup A: 10 W (5 patients) Subgroup B: 30 W (5 patients) Subgroup C: 50 W (5 patients)
  Interventions: Procedure: ex-vivo RFA under US control at 10 Watts (W) of power in 3 differents arms of lesions; Procedure: ex-vivo RFA under US control at 30 Watts (W) of power in 3 differents arms of lesions; Procedure: ex-vivo RFA under US control at 50 Watts (W) of power in 3 differents arms of lesions
- resected neuroendocrine tumors (Experimental): Subgroup A: 10 W (5 patients) Subgroup B: 30 W (5 patients) Subgroup C: 50 W (5 patients)
  Interventions: Procedure: ex-vivo RFA under US control at 10 Watts (W) of power in 3 differents arms of lesions; Procedure: ex-vivo RFA under US control at 30 Watts (W) of power in 3 differents arms of lesions; Procedure: ex-vivo RFA under US control at 50 Watts (W) of power in 3 differents arms of lesions

INTERVENTIONS:
Procedure: ex-vivo RFA under US control at 10 Watts (W) of power in 3 differents arms of lesions — 5 PDAC with neoadjuvant chemotherapy treated at 10 W with ex-vivo RFA 5 PDAC without previous neoadjuvant chemotherapy treated at 10 W with ex-vivo RFA 5 NET treated at 10 W with ex-vivo RFA
Procedure: ex-vivo RFA under US control at 30 Watts (W) of power in 3 differents arms of lesions — 5 PDAC with neoadjuvant chemotherapy 5 PDAC without previous neoadjuvant chemotherapy 5 NETs
Procedure: ex-vivo RFA under US control at 50 Watts (W) of power in 3 differents arms of lesions — 5 PDAC with neoadjuvant chemotherapy 5 PDAC without previous neoadjuvant chemotherapy 5 NETs

SUMMARY:
The study investigates the feasibility and the efficacy to treat pancreatic solid lesions as pancreatic adenocarcinomas (PDAC) and neuroendocrine tumors (NET) with ex-vivo radiofrequency ablation (RFA) under ultrasound (US) control.

The study intent is to define the optimal radiofrequency ablation POWER of the system in terms of maximum sizes (diameters) of histological coagulative necrosis obtained at pathological samples. Results will be useful to define the optimal settings to ablate pancreatic solid lesions (PDAC and neuroendocrine tumours).

DETAILED DESCRIPTION:
A probe specifically designed for Endoscopic Ultrasound (EUS) in vivo treatment of human pancreatic solid masses will be used. The probe is connected to a radiofrequency generator on which the power can be set and the tip of the probe (on the tip is present the radiofrequency electrode) is continuously perfused by chilled solution. The generator can stop the power supply when the tissue impedance goes beyond the threshold value to prevent tissue carbonization

ELIGIBILITY:
Inclusion Criteria: pancreatic solid lesion presence (pancreatic adenocarcinoma and neuroendocrine tumors) resected during pancreatic surgery -

Exclusion Criteria: no signature on informed consent

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-09-12 (Actual); Primary Completion 2020-06-12 (Actual); Study Completion 2020-06-12 (Actual)

PRIMARY OUTCOMES:
diameter (millimeters) of coagulative necrosis obtained by RadioFrequency Ablation | within 15-20 days
  assesses by two blinded pathologists

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS San Raffaele Hospital, Milan, Italy

IPD SHARING:
Plan to Share IPD: No